CLINICAL TRIAL: NCT01088763
Title: A PHASE 1/2 STUDY OF RO4929097, AN ORAL SMALL MOLECULE INHIBITOR OF GAMMA-SECRETASE, IN CHILDREN WITH RELAPSED/REFRACTORY SOLID OR CNS TUMORS, LYMPHOMA, OR T-CELL LEUKEMIA
Brief Title: Gamma-Secretase Inhibitor RO4929097 in Treating Young Patients With Relapsed or Refractory Solid Tumors, CNS Tumors, Lymphoma, or T-Cell Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02024; NCI-2011-02024 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ADVL0919; CDR0000667505; ADVL0919 (Other: Children's Oncology Group); ADVL0919 (Other: CTEP); U01CA097452 (NIH)
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2011-10

CONDITIONS: Childhood Atypical Teratoid/Rhabdoid Tumor; Childhood Central Nervous System Choriocarcinoma; Childhood Central Nervous System Germinoma; Childhood Central Nervous System Mixed Germ Cell Tumor; Childhood Central Nervous System Teratoma; Childhood Central Nervous System Yolk Sac Tumor; Childhood Choroid Plexus Tumor; Childhood Craniopharyngioma; Childhood Ependymoblastoma; Childhood Grade I Meningioma; Childhood Grade II Meningioma; Childhood Grade III Meningioma; Childhood Infratentorial Ependymoma; Childhood Medulloepithelioma; Childhood Mixed Glioma; Childhood Oligodendroglioma; Childhood Supratentorial Ependymoma; Gonadotroph Adenoma; Pituitary Basophilic Adenoma; Pituitary Chromophobe Adenoma; Pituitary Eosinophilic Adenoma; Prolactin Secreting Adenoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Central Nervous System Embryonal Tumor; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Ependymoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Medulloblastoma; Recurrent Childhood Pineoblastoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Childhood Spinal Cord Neoplasm; Recurrent Childhood Subependymal Giant Cell Astrocytoma; Recurrent Childhood Supratentorial Primitive Neuroectodermal Tumor; Recurrent Childhood Visual Pathway and Hypothalamic Glioma; Recurrent Childhood Visual Pathway Glioma; Recurrent Pituitary Tumor; Recurrent/Refractory Childhood Hodgkin Lymphoma; T-cell Childhood Acute Lymphoblastic Leukemia; T-cell Large Granular Lymphocyte Leukemia; TSH Secreting Adenoma; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Rhabdoid Tumor; Choroid Plexus Neoplasms; Oligodendroglioma; Adenoma, Basophil; Adenoma, Chromophobe; Adenoma, Acidophil; Prolactinoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic; Astrocytoma; Familial ependymoma; Dendritic Cell Sarcoma, Interdigitating; Medulloblastoma; Burkitt Lymphoma; Spinal Cord Neoplasms; Optic Nerve Glioma; Pituitary Neoplasms; Recurrence; Leukemia, Large Granular Lymphocytic | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide; Dexamethasone; Calcium Dobesilate

ARMS (1):
- Arm I (Experimental): GROUP A: Patients receive oral gamma-secretase inhibitor RO4929097 once daily on days 1-3, 8-10, 15-17, and 22-24. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  GROUP B: Patients receive oral gamma-secretase inhibitor RO4929097 once daily on days 1-5, 8-12, 15-19, and 22-26. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity. Patients may also receive concurrent oral dexamethasone twice daily on the days of gamma-secretase inhibitor RO4929097 administration.
  Once the MTD or recommended phase II dose of RO4929097 plus dexamethasone in children with solid tumors, including CNS tumors, or lymphoma has been identified, this dose is used for patients with relapsed-refractory T-ALL (phase 2 portion of the study) to evaluate RO4929097 in combination with dexamethasone using one of the studied schedules.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Other: diagnostic laboratory biomarker analysis; Other: pharmacological study; Drug: dexamethasone

INTERVENTIONS:
Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097 — Given PO
  Other Names: R4733; RO4929097
Other: diagnostic laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Drug: dexamethasone — Given IV
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM

SUMMARY:
This phase I/II clinical trial is studying the side effects and best dose of gamma-secretase inhibitor RO4929097 and to see how well it works in treating young patients with relapsed or refractory solid tumors, CNS tumors, lymphoma, or T-cell leukemia. Gamma-secretase inhibitor RO4929097 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum-tolerated dose (MTD) and recommend a phase II dose of gamma-secretase inhibitor RO4929097 administered orally to children with relapsed or refractory solid tumors or lymphoma on two schedules: once daily orally on a 3-day on/4-day off weekly schedule (schedule A) or once daily for 5 consecutive days weekly schedule (schedule B).

II. To define and describe the toxicities of this drug administered on these schedules to children with relapsed or refractory solid tumors, lymphoma, or T-cell leukemia.

III. To estimate the MTD and recommended phase II dose of gamma-secretase inhibitor RO4929097 administered with dexamethasone.

IV. To define and describe the toxicities of gamma-secretase inhibitor RO4929097 administered with dexamethasone.

V. To characterize the pharmacokinetics of gamma-secretase inhibitor RO4929097 in children with refractory cancer.

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of gamma-secretase inhibitor RO4929097 in children with solid or CNS tumors and lymphoma within the confines of a phase I study.

II. To obtain initial efficacy data on the antitumor activity of gamma-secretase inhibitor RO4929097 when combined with dexamethasone in children with relapsed-refractory T-cell leukemia (T-acute lymphoblastic leukemia [ALL]).

III. To study the effect of gamma-secretase inhibitor RO4929097 on Hes1 (hairy/enhancer of split) and other components of the Notch signaling pathway in peripheral blood mononuclear cells and/or T-ALL blasts. (exploratory) IV. To examine archival tumor samples for expression of JAGGED1, JAGGED2, cleaved NOTCH1, and HES1, and HES5 by IHC and for amplification of NOTCH1 or NOTCH2 using FISH analysis. (exploratory) V. To preliminarily assess changes following treatment with gamma-secretase inhibitor RO4929097 using FDG PET imaging. (exploratory)

OUTLINE: This is a multicenter, phase I, dose-escalation study of gamma-secretase inhibitor RO4929097 followed by a phase II study. Patients are enrolled sequentially to group A or B.

GROUP A: Patients receive oral gamma-secretase inhibitor RO4929097 once daily on days 1-3, 8-10, 15-17, and 22-24. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

GROUP B: Patients receive oral gamma-secretase inhibitor RO4929097 once daily on days 1-5, 8-12, 15-19, and 22-26. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity. Patients may also receive concurrent oral dexamethasone twice daily on the days of gamma-secretase inhibitor RO4929097 administration.

Once the MTD or recommended phase II dose of RO4929097 plus dexamethasone in children with solid tumors, including CNS tumors, or lymphoma has been identified, this dose is used for patients with relapsed-refractory T-ALL (phase 2 portion of the study) to evaluate RO4929097 in combination with dexamethasone using one of the studied schedules. Blood, plasma, bone marrow, and tumor tissue samples may be collected at baseline and periodically during the first course for correlative lab and tumor studies, including pharmacokinetics.

After completion of study treatment, patients are followed up for up to 30 days.

*NOTE: This trial was intended to be Phase I/II, but the trial never continued to the Phase II portion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy (at diagnosis or relapse)

  * Biopsy not required for intrinsic brain stem tumors or optic pathway gliomas
* No B-cell precursor acute lymphoblastic lymphoma (ALL) or acute myeloid leukemia
* No T-cell leukemia with CNS3 disease
* Measurable or evaluable disease
* Current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Neurologic deficits in patients with CNS tumors must have been relatively stable for 1 week
* No active CNS leukemia
* Karnofsky performance status (PS) 50-100% (for patients > 16 years of age) or Lansky PS 50-100% (for patients ≤ 16 years of age)

  * Patients who are unable to walk because of paralysis,but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the PS
* Patients with solid tumors without bone marrow involvement must meet the following criteria:

  * Peripheral ANC ≥ 1,000/mm^3
  * Platelet count ≥ 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions within the past 7 days)
  * Hemoglobin ≥ 8.0 g/dL (may receive RBC transfusions)
* Patients with known bone marrow metastatic disease must meet the above criteria and must not be known to be refractory to red cell or platelet transfusion
* Patients with leukemia must meet the following criteria:

  * Platelet count ≥ 20,000/mm^3 (may receive platelet transfusions)
  * Hemoglobin ≥ 8.0 g/dL (may receive RBC transfusions)
  * Must not be known to be refractory to RBC or platelet transfusions
* Creatinine clearance or radioisotope GFR ≥ 70 mL/min OR a serum creatinine based on age/gender as follows:

  * ≤ 0.6 mg/dL (patients 1 to < 2 years)
  * ≤ 0.8 mg/dL (patients 2 to < 6 years)
  * ≤ 1 mg/dL (patients 6 to < 10 years)
  * ≤ 1.2 mg/dL (patients 10 to < 13 years)
  * ≤ 1.4 mg/dL (female patients ≥ 13 years)
  * ≤ 1.5 mg/dL (male patients 13 to < 16 years)
  * ≤ 1.7 mg/dL (male patients ≥ 16 years)
* Bilirubin (sum of conjugated and unconjugated) ≤ 1.5 times upper limit of normal (ULN) for age
* ALT ≤ 110 U/L (for the purpose of this study, the ULN for ALT is 45 U/L)
* Serum albumin ≥ 2 g/dL
* No uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia, or hypokalemia defined as < lower limit of normal despite adequate electrolyte supplementation
* Baseline QTc < 450 msec
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception (i.e., one highly effective method and one additional effective method) for ≥ 4 weeks before, during, and for ≥ 12 months after completion of study treatment
* Female patients may not donate ova during or after study treatment
* Able to comply with the safety monitoring requirements of the study, in the opinion of the investigator
* Able to swallow tablets and capsules
* No known malabsorption syndrome or other condition that would interfere with intestinal absorption
* No known serological positivity for hepatitis A, B, or C, no known history of liver disease, and no other forms of hepatitis or cirrhosis
* No known HIV positivity
* No uncontrolled infection
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to gamma-secretase inhibitor RO4929097 or dexamethasone
* Patients may not donate blood during or for ≥ 12 months after completion of study treatment
* No hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia, or hypokalemia that is uncontrolled despite adequate electrolyte supplementation
* No prior gamma-secretase inhibitor RO4929097
* Fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy
* More than 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosourea) (for patients with solid tumors, CNS tumors, or lymphomas)
* Patients with T-cell leukemia must meet the following criteria:

  * Patients who relapsed on standard ALL maintenance chemotherapy must not have received maintenance chemotherapy within the past 3 days
  * Patients who relapsed when they were not receiving standard ALL maintenance therapy are eligible provided it has been ≥ 14 days since the completion of cytotoxic chemotherapy with the exception of hydroxyurea
  * Cytoreduction with hydroxyurea can be initiated and continued for up to 24 hours before the start of study treatment
* At least 6 months since prior total-body irradiation (TBI), craniospinal radiotherapy, or radiotherapy to ≥ 50% of the pelvis
* At least 6 weeks since other prior substantial bone marrow radiotherapy
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 3 months since prior stem cell transplantation or rescue without TBI and no evidence of active graft-vs-host disease
* At least 7 days since the completion of therapy with a biologic agent

  * For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur (the duration of this interval must be discussed with the study chair)
* At least 7 days or 3 half-lives, whichever is longer, since prior treatment with a monoclonal antibody
* More than 7 days since prior growth factors that support platelet or white cell number or function
* At least 7 days since prior corticosteroids
* No other concurrent investigational drugs
* No other concurrent anticancer agents including chemotherapy (except for hydroxyurea), radiotherapy, immunotherapy, or biologic therapy

  * Patients with T-ALL who benefit from treatment with gamma-secretase inhibitor RO4929097 in combination with dexamethasone may receive intrathecal methotrexate
* No concurrent warfarin sodium (Coumadin®)
* No concurrent medications that are strong inducers and/or inhibitors of CYP3A4
* No concurrent medications or food that may interfere with the metabolism or gamma-secretase inhibitor RO4929097, including ketoconazole and fresh-squeezed grapefruit juice

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 129 (Actual)
Dates: Start 2010-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of RO4929097 determined according to dose-limiting toxicities (DLTs) graded using Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0) | 28 days
MTD of RO4929097 administered with dexamethasone determined according to DLTs graded using CTCAE v4.0 | 28 days

SECONDARY OUTCOMES:
Antitumor activity of RO4929097 with or without dexamethasone assessed by Response Evaluation Criteria for Solid Tumors (RECIST) | Up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Najat Daw, Principal Investigator — Children's Oncology Group
Locations (12):
- United States (11):
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Stanford University Hospitals and Clinics, Stanford, California
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada